CLINICAL TRIAL: NCT04847505
Title: Pragmatic Study on the Use of 68Ga-DOTA-TATE PET|CT Imaging as a Standard of Care to Influence Clinical Management
Brief Title: 68Ga-DOTA-TATE PET/CT Imaging in NETs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, Head of the clinical research, CIMS, CHUS, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIMS-2019-02
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Neuroendocrine Tumors
Keywords: 68Ga-DOTA-TATE; PET imaging; Pragmatic study; Neuroendocrine tumors (NET)
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Neuroendocrine cancer patients, regardless of the primary tumor origin, are eligible. Recruitment is across all Canada but the examination is performed at the primary site of the study. The safety profile of the procedure will be assessed, and integration of 68Ga-DOTA-TATE will be integrated in the routine clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neuroendocrine cancer patients (Experimental): All neuroendocrine cancer patients referred by their physician and fulfilling the eligibility criteria across Canada can be recruited to the primary site of the study. Patients will be injected intravenously with 3 MBq/kg (maximum 370 MBq) of 68Ga-DOTA-TATE. 45-90 minutes following injection, patients will be imaged in a PET/CT scanner. Images will be analyzed by a trained nuclear medicine physician.
  Safety profile, eventual adverse effects, false positives, false negatives and any abnormal biodistribution of the radiotracer will be monitored and analysed.
  Interventions: Diagnostic Test: 68Ga-DOTA-TATE

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-TATE — The intervention consists of an intravenous injection of the radiopharmaceutical 68Ga-DOTA-TATE and a physiological saline flush, followed 45-90 minutes later by a PET/CT image acquisition.
  Other Names: Netspot

SUMMARY:
This clinical trial is a pragmatic study aiming to evaluate the innocuity/safety profile of the PET radiotracer 68Ga-DOTA-TATE, and to establish the procedure as a routine standard-of-care diagnostic tool for all neuro-endocrine cancer patients. It is a single-center study, but with recruitment across all Canada. The trial is prospective, non-randomized, open-label and with no control group. The superiority of this procedure over the former standard-of-care (Octreoscan) was already established in previous and numerous studies across the world. As such, the current trial aims to gather data to further support the implementation of 68Ga-DOTA-TATE as the new standard-of-care for neuro-endocrine tumors (NET).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical requisition for a 68Ga-DOTA-TATE PET/CT signed by a referring doctor
2. Patients with suspected or proven tumors expressing somatostatin receptors
3. Informed consent by patient (or parents if patient is less than 18 years of age)

Exclusion Criteria:

1. *Pregnancy (not an absolute exclusion). See below*.
2. Patient refusal to participate.
3. Prior severe anaphylactic reaction to DOTA-TATE or somatostatin analogs.

   * In the case of a diagnostic procedure in a patient who is or may be pregnant, the principle of benefits-disadvantages would be applied following an in-depth discussion with the treating physicians and the patient. In this context, any clinical situation in which the patient's life would be at stake by excluding her from the study would be considered. The conditions to decide whether to include the patient would be:

     * Severe medical condition involving the life of the pregnant woman and/or the fetus;
     * Existing treatments that are ineffective or may present toxicity to the woman and/or fetus;
     * High clinical suspicion of a somatostatin receptor overexpressing tumour;
     * Negative, indeterminate or contraindicated first-line imaging tests;
     * Therapeutic gesture considered during pregnancy based on the results of the examination, which may include termination of pregnancy or premature delivery;
     * Documented discussion with the treating team and the patient;
     * Patient agrees.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety profile of 68Ga-DOTA-TATE | 5 years
  Following the injection, the patient will be explicitly reminded of possible symptoms and undesirable events. The patient will be advised to inform the study personnel of the occurrence of any events, at the most opportune time. The patient will be instructed to call the local nuclear medicine study coordinator for any undesirable event that may occur for 48 hours after the PET/CT scan.
  Safety will be assessed by compiling all reported adverse events. Adverse events reported by patients or observed by the investigator will be recorded in the patients' CRFs, the AE database, and reported to the research manager.

SECONDARY OUTCOMES:
Generate clinical information on the impact of 68Ga-DOTA-TATE for NET patient management | 5 years
  Neuroendocrine tumors (NET) used to be difficult to diagnose early with conventional methods, but with the advent of new-generation Somatostatin Receptor radioligands such as 68Ga-DOTA-TATE precise and early detection is now frequent. This trial offers the opportunity to evaluate the impact of this state-of-the-art diagnostic procedure on the management of NET patients on a large, nation-wide cohort. As such, the research team will monitor the clinical gain of 68Ga-DOTA-TATE on the diagnostic and management of NETs regarding sensitivity, specificity and accuracy compared to previous diagnostic methods.
Instigate the routine standard-of-care use of 68Ga-DOTA-TATE for NET patients | 5 years
  Clinical and scientific evidences showed that 68Ga-DOTA-TATE is vastly superior as a diagnostic tool than the current standard-of-care Octreoscan. As such, this trial aims to implement 68Ga-DOTA-TATE as the new standard-of-care for precision diagnostic of NETs. In order to do so, health policy agencies (most notably Health Canada) will be notified about the gains (or the flaws if any) of 68Ga-DOTA-TATE over the current standard-of-care (Octreoscan) for the precise diagnostic and follow-up of NETs that will be observed during the present study. The safety profile and diagnostic accuracy assessed in Outcome 1 and 2 will be used to convince the authorities of the net benefit of using this procedure rather than the "old" standard-of-care.

CONTACTS AND LOCATIONS:
Overall Officials: Éric E Turcotte, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (2):
- Canada (2):
  - Centre Intégré Universitaire de Santé et des Services Sociaux du Centre de l'Ouest de Montréal - Jewish General Hospital, Montreal, Quebec
  - CHUS, Sherbrooke, Quebec